CLINICAL TRIAL: NCT04664335
Title: Impact of Endometriosis on Pregnancy and Delivery - a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. med. Sebastian Daniel Schäfer, Head of Gynecology, University Hospital Muenster
Other Study IDs: Schäfer_Endo_Preg_Del_Comp
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Endometriosis; Pregnancy Complications; Delivery Complication; Complication; Miscarriage
Keywords: endometriosis; pregnancy; delivery; miscarriage; cesarian section
MeSH Terms: conditions — Endometriosis; Pregnancy Complications; Abortion, Spontaneous | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometriosis cases: endometriosis laparoscopically removed / child wish
  Interventions: Other: questionnaire
- controls: endometriosis laparoscopically excluded / child wish
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — if no Reply to questionnaire, telephone interview
  Other Names: interview

SUMMARY:
Purpose:

To study the impact of endometriosis on subsequent pregnancy and delivery.

Methods:

retrospective analysis by questionnaire / interview of cases (endometriosis laparoscopically removed / child wish) vs. controls (endometriosis laparoscopically excluded / child wish) from the University Hospital Muenster, Germany, treated between 2009 and 2016; analysis of pregnancy rate, mode of delivery and complications using Clavien-Dindo-classification, role of deep infiltrating endometriosis using ENZIAN classification; data analysis using t-test with p < 0.050% being considered significant.

ELIGIBILITY:
Inclusion Criteria:

* cases: Operation because of endometriosis at the endometriosis Center, University Hospital Muenster, child wish, wants to participate, correct age group
* controls: Operation because of sterility, exclusion of endometriosis during this Operation, child wish, wants to participate, correct age group

Exclusion Criteria:

* cases / controls: declines participation, incorrect age Group, no child wish

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: cases (endometriosis laparoscopically removed / child wish) vs. controls (endometriosis laparoscopically excluded / child wish) from the University Hospital Muenster, Germany, treated between 2009 and 2016
Sampling Method: Probability Sample
Enrollment: 1762 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | through study completion, an average of 1 year
  pregnancy rate
complications | through study completion, an average of 1 year
  complications during pregnancy, delivery, puerperium

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian D Schaefer, MD PhD, Principal Investigator — University Hospital Muenster, Germany
Locations (1):
- University Hospital Münster Germany, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
will share upon reasonable request according to regulations